CLINICAL TRIAL: NCT04506684
Title: Reveal LINQ Respiration Clinical Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20022
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Rate
Keywords: Reveal LINQ device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Investigational RAMware downloaded onto Reveal LINQ device — The study is utilizing an investigational RAMware, either LINQ HF or ALLEVIATE-HF, that will be downloaded onto the subject's market-released Medtronic Reveal LINQ ICM. The investigational RAMware enables the hardware to record and store additional sensor data from which a respiratory rate will be derived.

SUMMARY:
The LINQ™ Respiration study will collect and characterize Reveal LINQ™ derived respiration data from patients undergoing a simulated 24-hour time period while being monitored with capnography.

DETAILED DESCRIPTION:
The Reveal LINQ™ Respiration study is a Non-Significant Risk IDE, observational, non-randomized, multi-center, clinical study. The study is expected to be conducted at up to 5 centers in the United States and up to 100 subjects will be enrolled, with no more than 25 subjects enrolled per site. In addition, a minimum of 30% of all enrolled subjects will have a history of heart failure.

All enrolled subjects will either have the investigational LINQ HF or ALLEVIATE-HF RAMware downloaded onto their implanted Reveal LINQ device, Holter monitor and capnography monitor applied and undergo a series of activity and breathing maneuvers. The expected duration of subject participation in the study (from start of study procedures to study exit) is approximately 1.5 hours. The expected total study duration (from time of first enrollment to the exit of last enrolled subject) is approximately 3 months.

All Adverse events will be collected throughout the study duration of a subject's participation in the study, beginning at the time of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 55 years old
* Patient (or patient's legally authorized representative) is willing and able to provide written informed consent
* Patient is willing and able to comply with the study procedures
* Patient has an active Medtronic Reveal LINQ device that has been implanted for ≥ 60 days and no more than 3 years

Exclusion Criteria:

* Patient has an existing condition that necessitates the use of supplemental oxygen
* Patient has an active acute respiratory infection or a respiratory disorder that may affect ability to perform respiratory maneuvers
* Patient has NYHA Class IV heart failure per most recent assessment
* Any concomitant condition that might endanger the patient through participation in the study or interfere with study procedures, as assessed by the investigator
* Patient is enrolled in another study that could confound the results of this study
* Patient has an existing implantation of Medtronic IPG, ICD, CRT-D or CRT-P device

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population for the LINQ Respiration study will include subjects who are ≥ 55 years old and implanted with a Reveal LINQ device for ≥60 days and no longer than 3 years. In addition, a minimum of 30% of all enrolled subjects will have a documented history of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Demonstrating an agreement between LINQ and capnography derived respiratory rate | 6 months
  The primary objective is to demonstrate an acceptable agreement between Reveal LINQ™ derived respiratory rate and capnography waveform-derived respiratory rate.

SECONDARY OUTCOMES:
Characterizing the agreement between LINQ and capnography derived respiratory rate | 6 months
  The secondary objective is to characterize the agreement between Reveal LINQ™ derived respiratory rate with capnography waveform-derived respiratory rate utilizing all paired measurements captured during the study protocol.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cardiac Arrhythmia Service, Boca Raton, Florida
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - The Stern Cardiovascular Foundation, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD